CLINICAL TRIAL: NCT00672906
Title: Group Parent Training for Adolescent Eating Disorders
Acronym: GPT-AN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00010889; 5K23MH070418-03 (NIH); 7767 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-05

CONDITIONS: Adolescent Anorexia Nervosa; Subthreshold Anorexia Nervosa
Keywords: anorexia nervosa; group parent training; caregiver burden; eating disorders; treatment
MeSH Terms: conditions — Anorexia Nervosa; Caregiver Burden; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group Parent Training/Adolescent Skills Training
  Interventions: Behavioral: Group Parent Training
- Active Comparator (Active Comparator): Family Therapy according to the Maudsley Model
  Interventions: Behavioral: Maudsley Family Therapy

INTERVENTIONS:
Behavioral: Group Parent Training — Skills group for parents that provides psychoeducation for eating disorder and skills in behavior management, self-regulation, and emotion regulation.
  Arms: 1
Behavioral: Maudsley Family Therapy — Family therapy specifically adapted for the treatment of adolescent anorexia nervosa.
  Arms: Active Comparator

SUMMARY:
While parents are considered essential for the effective treatment of adolescents with anorexia nervosa, the most effective manner to involve parents in treatment is unknown. Given reports of high caregiver burden among parents of this clinical group, finding treatments that minimize parent burden while improving the child's eating disorder symptoms is essential.

This investigation will examine the preliminary effectiveness of a parent skills group and adolescent skills group compared to family therapy for the treatment of adolescent anorexia nervosa. The target of this intervention is the improvement of eating disorder symptoms in the child and improving self-efficacy, emotion regulation, and perceived burden in the parent.

The effectiveness of this experimental treatment group (Group Parent Training for the parents/Adolescent Skills Training for the adolescent) will be compared to the Maudsley model of family therapy. The effectiveness of the group program will be examined by exploring changes within individuals over time as well as via comparisons across treatment conditions. Results from this investigation will be used to calculate treatment effect sizes in the design of a larger, fully powered, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* age 11-18 years old
* living at home
* meet criteria for anorexia nervosa or subthreshold anorexia nervosa

Exclusion Criteria:

* no active psychosis
* no current suicidality
* medically safe for outpatient treatment

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2005-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 12 months

SECONDARY OUTCOMES:
Eating disorder symptoms other than body weight. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States